CLINICAL TRIAL: NCT01940705
Title: A Simplified Patient Centered Educational Tool for Improved Hearing Aid Outcomes
Brief Title: A Simplified Patient-Centered Educational Tool for Improved Hearing-Aid Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1260-R; 1I01RX001260-01 (NIH); 3224 (Other: Portland VA IRB)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Hearing Loss
Keywords: hearing aids; counseling; outcomes assessment (health care); rehabilitation
MeSH Terms: conditions — Hearing Loss | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard of care (SoC) (Active Comparator): standard of care hearing-aid orientation as provided by clinical audiologist
  Interventions: Other: Standard of Care
- SoC plus hearing-aid informational guide (Experimental): standard of care hearing-aid orientation as provided by clinical audiologist plus a take-home informational guide regarding their hearing aids
  Interventions: Other: Hearing-Aid Informational Guide; Other: Standard of Care
- SoC plus hearing aid DVD (Experimental): SoC hearing-aid orientation as provided by clinical audiologist plus a take-home hearing aid digital video disc
  Interventions: Other: Hearing-Aid DVD; Other: Standard of Care
- Soc plus teach-back technique (Experimental): standard of care hearing-aid orientation as provided by clinical audiologist plus a teach-back technique session reviewing information on the hearing aids
  Interventions: Behavioral: Teach-back Technique; Other: Standard of Care

INTERVENTIONS:
Other: Hearing-Aid Informational Guide — Printed take-home guide on hearing aids
  Arms: SoC plus hearing-aid informational guide
Other: Hearing-Aid DVD — Take-home DVD about hearing aids
  Arms: SoC plus hearing aid DVD
Behavioral: Teach-back Technique — Counseling/Educational session using the teach-back technique to review information about their hearing aids
  Arms: Soc plus teach-back technique
Other: Standard of Care — standard of care hearing-aid orientation as provided by clinical audiologist

SUMMARY:
Hearing loss is the second most prevalent service-connected disability among Veterans. Hearing aids are the most common technological intervention for hearing loss. The VA, therefore, spends a considerable amount of money on them. Despite these expenditures, there are some Veterans who do not use their hearing aids successfully. Research has demonstrated that this inconsistent use may be related to a patient's inability to effectively take care of, and use, hearing aids. The proposed investigation will compare the effectiveness of three different tools for enhancing the educational efforts (hearing-aid orientation) typically provided by clinical audiologists when dispensing hearing aids. Each of these educational tools were developed using established methods for improving patient-provider communication. The investigators hypothesize that the use of these tools will result in better hearing-aid outcomes for Veteran patients than using the current standard-of-care procedures.

DETAILED DESCRIPTION:
Objectives: Reasons for non-use of hearing aids are varied, but many studies have suggested that a lack of knowledge about how to use and/or take care of the hearing aids is a major factor. This is not surprising given that other healthcare fields have reported that between 40-80% of information provided during a clinical appointment is forgotten by the patient immediately after the appointment and almost half of what is remembered is not correct. The long-term goal of this project is to improve the delivery of information during the hearing-aid orientation, as better delivery of information will result in better hearing-aid handling skills and thus better overall hearing-aid outcomes. To accomplish this goal, the investigators propose to refine and evaluate the effectiveness of three forms of supplemental hearing-aid-orientation tools, each of which was developed using established guidelines for good patient-provider communication.

Plan: The purpose of the proposed application is to evaluate the relative effectiveness of four forms of hearing-aid orientation provided to first time hearing-aid users, three of which use some of the aforementioned strategies to enhance the standard of care. The four forms of orientation will be: (1) the standard-of-care hearing-aid orientation; (2) the standard of care plus provision a hearing-aid information guide (HAIG) (3) the standard of care supplemented by an explanation of its content using the talk-back technique to confirm patient understanding; and (4) the standard of care plus provision of a take-home hearing-aid orientation DVD (HAO DVD). The content of the HAIG will be field tested and finalized following input obtained via focus groups with clinical audiologists and first-time hearing aid users.

Methods: For the field testing up to 16 clinical audiologists and 10 new hearing aid user Veterans will be recruited to participate in focus groups during which they will view and then be asked questions about the content of the HAIG. Information learned during these focus groups will then be incorporated into the HAIG, at which time they will be ready for use in the study. For the comparative effectiveness study, up to 468 hearing-impaired Veterans who are about to become first-time hearing-aid users will be enrolled to participate in this investigation. These individuals will be recruited from the VA Portland Health Care System's Audiology and Speech Pathology Service (ASPS). Prior to receiving their hearing aids, subjects will be enrolled in the study at the National Center for Rehabilitative Auditory Research (NCRAR), and will conduct health literacy, manual dexterity and hepatic sensitivity, visual acuity, and learning and memory assessments. They will then attend their hearing aid fitting in the ASPS and will receive standard-of-care hearing-aid orientation. At the end of that appointment, they will receive one of the four study interventions. Subjects will return to the NCRAR 4-6 weeks after the hearing-aid-fitting appointment to complete the following outcome measures: a knowledge and practical test regarding hearing-aid use and care, a measure of self-efficacy, and a measure of hearing-aid outcomes. They also will be interviewed so that the investigators can learn their opinions about the intervention. A subset of the initial 50 participants enrolled into each study arm will attend a second follow-up appointment 6 months after the fitting appointment so the investigators can examine longer-term impacts of the hearing aid orientation interventions.

ELIGIBILITY:
Inclusion Criteria:

Participants will be Veterans who are receiving hearing aids from the Audiology Clinic at the VA Portland Health Care System and who have had no prior experience using hearing aids. To be included in the study, participants will:

* Be approved and have plans to get bilateral hearing aid fitting at the VA Portland Health Care System .
* Be able to read and converse in English.

Exclusion Criteria:

* Be younger than 50 years or older than 89 years of age.
* Have a documented diagnosis of neurological, cognitive, visual, or other mental disorder, such as Alzheimer's disease, schizophrenia, current alcohol or substance abuse, as determined by chart review that would interfere with study completion.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Samantha Lewis, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR; Gabrielle H Saunders, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Plus Hearing-aid Informational Guide: standard of care hearing-aid orientation as provided by clinical audiologist plus a take-home informational guide regarding their hearing aids
  Hearing-Aid Informational Guide: Printed take-home guide on hearing aids
  Standard of Care: standard of care hearing-aid orientation as provided by clinical audiologist
- Standard of Care Plus a Take-home Digital Video Disc: standard of care hearing-aid orientation as provided by clinical audiologist plus a take-home digital video disc regarding hearing aids
  Hearing-Aid digital video disc : Take-home digital video disc about hearing aids
  Standard of Care: standard of care hearing-aid orientation as provided by clinical audiologist
- Standard of Care Plus Counseling With the Teach-back Technique: standard of care hearing-aid orientation as provided by clinical audiologist plus a teach-back technique counseling session reviewing information on the hearing aids
  Teach-back Technique: Counseling/Educational session using the teach-back technique to review information about their hearing aids
  Standard of Care: standard of care hearing-aid orientation as provided by clinical audiologist
Period: Overall Study
Arm/Group | Standard of Care | Standard of Care Plus Hearing-aid Informational Guide | Standard of Care Plus a Take-home Digital Video Disc | Standard of Care Plus Counseling With the Teach-back Technique
Started | 66 | 67 | 69 | 67
Completed | 62 | 59 | 61 | 63
Not Completed | 4 | 8 | 8 | 4
Not completed — Lost to Follow-up | 1 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 2
Not completed — Intervention not given | 0 | 3 | 3 | 0
Not completed — Withdrawal by team - hearing aid change | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SoC Plus a Take-home DVD: standard of care hearing-aid orientation as provided by clinical audiologist plus a take-home DVD regarding hearing aids
  Hearing-Aid DVD: Take-home DVD about hearing aids
  Standard of Care: standard of care hearing-aid orientation as provided by clinical audiologist
- SoC Plus Counseling With the Teach-back Technique: standard of care hearing-aid orientation as provided by clinical audiologist plus a teach-back technique counseling session reviewing information on the hearing aids
  Teach-back Technique: Counseling/Educational session using the teach-back technique to review information about their hearing aids
  Standard of Care: standard of care hearing-aid orientation as provided by clinical audiologist
- Total: Total of all reporting groups
Arm/Group | Standard of Care | SoC Plus Hearing-aid Informational Guide | SoC Plus a Take-home DVD | SoC Plus Counseling With the Teach-back Technique | Total
Number analyzed (Participants) | 66 | 67 | 69 | 67 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (6.7) | 68.7 (7.6) | 69.3 (6.4) | 68.8 (7.0) | 69.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 5
  Male | 64 | 66 | 68 | 66 | 264
Region of Enrollment [Number; unit: participants]
  United States | 66 | 67 | 69 | 67 | 269

OUTCOME MEASURES:

1. Primary Outcome: Hearing Aid Skills and Knowledge Test
Description: Hearing Aid Skills and Knowledge measures knowledge and skills for tasks associated with hearing aid management, such as knowledge of and ability to change batteries, insert the hearing aid, etc. For knowledge scale, participant gives a verbal response. Items are assigned points: 0 (incorrect response) or 1 (correct response). For skills scale, participant conducts the required task. Items are assigned points: 0 (Could not perform task), 1 (Achieved with some difficulty, more than one attempt) or 2 (Achieved with no difficulty on first attempt).
  There were 15 knowledge items and 19 skill items. Percent correct was computed for each scale separately. Points were totaled, divided by the no. items with valid data, and multiplied by 100, with a correction to equate subscales.
  For the skills scale, percent correct scores were calculated based upon the notion that a value of 2 was considered 100% correct, 1 was considered 50% correct.
Time Frame: 4 weeks after the hearing-aid fitting
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- Standard of Care Plus a Take-home Digital Video Disc: standard of care hearing-aid orientation as provided by clinical audiologist plus a take-home DVD regarding hearing aids
  Hearing-Aid digital video disc: Take-home digital video disc about hearing aids
  Standard of Care: standard of care hearing-aid orientation as provided by clinical audiologist
Arm/Group | Standard of Care | Standard of Care Plus Hearing-aid Informational Guide | Standard of Care Plus a Take-home Digital Video Disc | Standard of Care Plus Counseling With the Teach-back Technique
Number analyzed (Participants) | 62 | 59 | 61 | 63
percentage of correct responses
  Hearing Aid Skills and Knowledge Test Knowledge | 65.4 (12.2) | 68.3 (12.3) | 66.2 (11.8) | 74.6 (12.3)
  Hearing Aid Skills and Knowledge Test Skill | 77.3 (11.2) | 80.3 (10.7) | 78.9 (9.4) | 83.0 (10.2)
Statistical Analysis 1: Comparison: Standard of Care vs Standard of Care Plus Hearing-aid Informational Guide vs Standard of Care Plus a Take-home Digital Video Disc vs Standard of Care Plus Counseling With the Teach-back Technique; Analysis for Hearing Aid Skills and Knowledge test Skills scale; Test type: Superiority; p = 0.001, ANOVA; Mean Difference (Final Values) = 5.578
Statistical Analysis 2: Comparison: Standard of Care vs Standard of Care Plus Hearing-aid Informational Guide vs Standard of Care Plus a Take-home Digital Video Disc vs Standard of Care Plus Counseling With the Teach-back Technique; Analysis for Hearing Aid Skills and Knowledge test Knowledge scale; Test type: Superiority; p = 0.003, ANOVA; Mean Difference (Final Values) = 4.235

2. Secondary Outcome: The Measure of Audiologic Rehabilitation Self-Efficacy for Hearing Aids
Description: 12-item questionnaire assessing self-efficacy for basic and advanced hearing aid handling skills. Item responses are on a scale of 0 to 100 in 10 point increments. Score of 0 = no self efficacy to100 = complete self efficacy. Final score is an average of individual item responses.
Time Frame: 4 weeks after the hearing-aid fitting
Population: Questionnaire data are missing due to a technical issue for one individual in the SoC plus hearing-aid informational guide arm and one in the SoC plus counseling with the teach-back technique
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | SoC Plus Hearing-aid Informational Guide | SoC Plus a Take-home DVD | SoC Plus Counseling With the Teach-back Technique
Number analyzed (Participants) | 62 | 58 | 61 | 62
units on a scale | 77.1 (15.3) | 78.4 (11.5) | 80.1 (12.4) | 80.9 (14.4)
Statistical Analysis 1: Comparison: Standard of Care vs SoC Plus Hearing-aid Informational Guide vs SoC Plus a Take-home DVD vs SoC Plus Counseling With the Teach-back Technique; Test type: Superiority; p = 0.414, ANOVA; Mean Difference (Final Values) = 0.956

3. Secondary Outcome: International Outcome Inventory for Hearing Aids.
Description: Hearing-aid outcomes questionnaire assessing benefit, satisfaction, use, etc. Seven items, each on a scale of 1-5. 1 = low satisfaction/benefit/use etc., 5 = maximum satisfaction/benefit/use etc. A total score is derived by summing the score from each of the seven items. Total scores range from a low of 7 to a high of 35.
Time Frame: 4 weeks after the hearing-aid fitting
Population: Questionnaire data are missing for one individual in the Standard of care arm, five in the SoC plus hearing-aid informational guide arm, five in the Standard of care plus a take-home digital video disc and two in the SoC plus counseling with the teach-back technique due to technical issues.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Standard of Care Plus Hearing-aid Informational Guide | Standard of Care Plus a Take-home Digital Video Disc | Standard of Care Plus Counseling With the Teach-back Technique
Number analyzed (Participants) | 61 | 54 | 56 | 61
units on a scale | 29.3 (4.2) | 29.7 (4.5) | 29.7 (4.1) | 30.0 (4.0)
Statistical Analysis 1: Comparison: Standard of Care vs Standard of Care Plus Hearing-aid Informational Guide vs Standard of Care Plus a Take-home Digital Video Disc vs Standard of Care Plus Counseling With the Teach-back Technique; Test type: Superiority; p = 0.847, ANOVA; Mean Difference (Final Values) = 0.270

ADVERSE EVENTS:
Arm/Group | Standard of Care | SoC Plus Hearing-aid Informational Guide | SoC Plus a Take-home DVD | SoC Plus Counseling With the Teach-back Technique
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/59 | 0/61 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/62 | 1/59 | 0/61 | 0/63
Other Adverse Events (participants affected / at risk) | 0/62 | 0/59 | 0/61 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=62) | SoC Plus Hearing-aid Informational Guide (N=59) | SoC Plus a Take-home DVD (N=61) | SoC Plus Counseling With the Teach-back Technique (N=63)
Non-study-related adverse event (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — During testing when participant removed right hearing aid, the research audiologist noted the dome was missing. Otoscopy revealed the dome was stuck in the ear canal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No